CLINICAL TRIAL: NCT00398203
Title: Safety and Efficacy of Using NaviAid™ BGE Device (Balloon Guided Endoscopy) For Endoscopic Diagnosis and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smart Medical Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLI-10111
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Intestinal Diseases
Keywords: NaviAid™ BGE Device; Small Intestine; Intestinal Diseases
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NaviAid™ BGE Device — NaviAid™ Balloon Guided Endoscopy Device
  Other Names: NaviAid™ Balloon Guided Endoscopy Device

SUMMARY:
To assess the efficacy of the NaviAid™ BGE Device, while used in conjunction with a standard endoscope for the diagnosis and treatment of the small intestine.

DETAILED DESCRIPTION:
Smart Medical Systems has developed the NaviAid™ Balloon Guided Endoscopy (BGE) Device, an innovative medical device for the GI tract diagnosis and treatment. The Balloon Guided Endoscopy (BGE) is a procedure intended for the examination of the small intestine, which utilizes the NaviAid™ BGE Device in conjunction with a standard endoscope.

The objectives of this prospective controlled study are to evaluate the safety and efficacy of using the NaviAid™ BGE device in the examination of the small intestine in conjunction with a standard endoscope.

Efficacy will be assessed by comparing NaviAid™ BGE Device performances to a reference Enteroscopy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female aged between 18-80 years (inclusive).
* Subject is scheduled for endoscopic procedure after the case was reviewed by one of the investigators.
* Symptomatic subject defined as having at least one of the following signs or symptoms:

  * Abdominal pain
  * Cramps
  * Bloating
  * Diarrhea
  * Nausea
  * Vomiting
  * Unexplained Anemia
  * GI bleeding from an unknown source
  * Small bowel abnormality on any imaging study
* Subject able to comprehend and give informed consent for participation in this study
* Signed Informed Consent Form

Exclusion Criteria:

* Pregnancy
* Acute bowel obstruction
* Concomitant Coumadin or warfarin use
* Severe diverticulitis
* Recent (within the last 3 months) coronary ischemia or CVA (stroke)
* Any chronic unstable disease
* Bleeding disorders
* Needing emergency surgery
* Any patient condition deemed too risky for SBE by the investigator
* Known cognitive or psychiatric disorder
* Physician objection
* Concurrent participation in any other clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy will be assessed by comparing NaviAid™ BGE Device performances to a reference Enteroscopy procedure in terms of depth of small intestine advancement and visualization. | Within 6 months of completion of the trial

SECONDARY OUTCOMES:
Safety of the NaviAid™ BGE Device will be assessed by reporting adverse events, and by comparing to a reference Enteroscopy procedure. | Within 6 months of completion of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Ingvar Bjarnason, Prof., Principal Investigator — Kings College Hospital
Locations (1):
- Kings College Hospital, London, United Kingdom